CLINICAL TRIAL: NCT03387267
Title: A Prospective Multi-center Study Comparing the Performance of the Dysphagia Detection System (DDS) in Detecting Impaired Swallowing Safety and Efficiency as Compared to the Clinical Reference Method - Videofluoroscopic Swallowing Study
Brief Title: Videofluoroscopic Swallowing Study (VFSS)
Acronym: PORSCHE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to futility
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Cytel Inc. (Industry); Regulatory and Clinical Research Institute Inc (Other); Nestec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 16.21.CLI
Record Dates: First submitted 2017-10-30; First posted 2018-01-02 (Actual); Results first posted 2021-05-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Parkinson Disease; Multiple Sclerosis; Oropharyngeal Dysphagia; Alzheimer Disease; Dementia
MeSH Terms: conditions — Stroke; Parkinson Disease; Multiple Sclerosis; Deglutition Disorders; Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: The clinical trial will initially start as a 3-look group sequential design (GSD). Alpha-spending will be calculated using Lan-DeMets spending function (with O'Brien-Fleming parameter). At the first interim analysis (IA-1) the threshold on the ROC curve may be re-computed using the ROC curve generated using the IA-1 data, in which case, the validation trial would start afresh following IA-1 using a 2-look GSD. Data included in the IA-1 would no longer be used for the validation phase.
Masking Description: An operationally seamless single-arm, prospective, multicenter, single-blinded for central outcomes assessors trial to test DDS in assessing swallowing safety and efficiency in patients at risk of oropharyngeal dysphagia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- single-arm Dysphagia Detection System (Other): An operationally seamless single-arm, prospective, multicenter, single-blinded for central outcomes assessors trial to test DDS in assessing swallowing safety and efficiency in patients at risk of oropharyngeal dysphagia.
  Interventions: Device: Dysphagia Detection System

INTERVENTIONS:
Device: Dysphagia Detection System — The Nestle Health Sciences (NHSc) Dysphagia Detection System (DDS) is a portable, non-invasive device designed for use at the bedside. The investigational DDS has 3 basic components: Sensor Unit (suspended on a necklace), Sensor Fixation and a personal computer (PC) for collecting data. The Sensor Unit consists of a dual-axis accelerometer in a plastic housing that is attached to the front of a patient's neck just below the thyroid cartilage by the single-use, disposable fixation unit. The Sensor Unit is connected via a cable to an A/D converter which then connects via cable to the PC. The PC collects the examination data, which is then sent to dedicated application software (installed at the CRO), which interprets the acceleration data and displays the examination result.

SUMMARY:
The study procedure of simultaneous VFSS and DDS measurement will be completed in one day and the subject will be followed within 2 business days after the study procedure to monitor for adverse events.

DETAILED DESCRIPTION:
DDS signals and VFSS will be recorded simultaneously (for the same bolus) using barium contrast agent stimuli prepared in three consistencies: thin, mildly-thick and moderately-thick. Subjects will undergo VFSS with simultaneous DDS using up to 5 boluses of thin barium stimulus ("THIN-Ba"), and up to 4 boluses of barium thickened to mildly ("MILD-Ba") thick and up to 4 boluses of moderately ("MODERATE-Ba") thick barium consistencies using Resource Thicken Up Clear Nestlé Health Science (TUC). 4, 3 and 3 boluses for THIN-Ba, MILD-Ba and MOD-Ba will be analyzed using the classifier algorithms for sensitivity/specificity results. According to the exploratory trial, VFSS data for safety or efficiency can be missing for up to 14% boluses due to quality of VFSS recording. To compensate for potential losses of boluses due to missing gold standard (VFSS) data, 5, 4 and 4 boluses will be collected for the three consistencies respectively . The DDS signals will be sent to a dedicated application software installed at the CRO, which interprets the acceleration data and displays the examination result. The VFSS recording will be sent to CRO and provided for blinded assessment by the independent central VFSS laboratory.The study procedure of simultaneous VFSS and DDS measurement will be completed in one day and the subject will be followed within 2 business days after the study procedure to monitor for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (over 18 years of age)
* Hospitalized subjects or outpatients identified as at risk of oropharyngeal dysphagia (using local practice)
* Patients belong to one of the following groups:

  * Stroke patients
  * Traumatic brain injury
  * Parkinson Disease (PD) stage III or higher by Hoehn and Yahr scale
  * Multiple Sclerosis (MS) above age 60
  * Alzheimer Disease (AD) or other Dementia
* Other medically complex hospitalized subjects not covered by the exclusion criteria and identified as at risk of dysphagia
* Subject is able to comply with VFSS protocol to diagnose dysphagia
* Subject is able to give voluntary, written informed consent to participate in the clinical investigation and from whom consent has been obtained / or a consultee has consented on he subjects behalf in line with nationally agreed guidelines concerning adults unable to consent for themselves.

Exclusion Criteria:

* Presence of nasogastric / nasojejunal feeding tube at the time of VFSS test
* Currently has a tracheostomy, or has had a tracheostomy in the past year
* Had posterior cervical spine surgery and/or carotid endarterectomy in the last 6 months
* Had significant surgery to the mouth and/or neck, for example resection for oral or pharyngeal cancer, radical neck dissection, anterior cervical spine surgery, orofacial reconstruction, pharyngoplasty, or thyroidectomy. Routine tonsillectomy and/or adenoidectomy are not excluded
* Experienced non-surgical trauma to the neck (e.g., knife wound) resulting in musculoskeletal or nerve injury in the neck.
* Received radiation or chemotherapy to the oropharynx or neck for cancer.
* Allergy to oral radiographic contrast media (specifically barium)
* Distorted oropharyngeal anatomy (e.g. pharyngeal pouch)
* Cognitive impairment that prevents them from being able to comply with study instructions and procedures
* Known to be pregnant at the time of enrollment
* Currently has significant facial hair at the location of sensor adherence and are unwilling/unable to be shaved
* Any patients the local investigator finds that participation would not be in patients' best interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Muhlemann, MD, Study Director — Nestle Health Science; Richard Harvey, MD, Principal Investigator — Shirley Ryan AbilityLab (Rehabilitation Institute of Chicago)
Locations (13):
- United States (12):
  - Rancho Research Institute, Rancho Los Amigos National Rehabilitation Center, Downey, California
  - University of Colorado Denver, Aurora, Colorado
  - Medstar Rehabilitation Hospital, Washington D.C., District of Columbia
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Marionjoy Rehabilitation Hospital, Wheaton, Illinois
  - Kentucky Clinic, Lexington, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - New York Presbyterian/Weill Cornell Medical Center, New York, New York
  - New York Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - The Burke Medical Research Institute, White Plains, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clave P, Shaker R. Dysphagia: current reality and scope of the problem. Nat Rev Gastroenterol Hepatol. 2015 May;12(5):259-70. doi: 10.1038/nrgastro.2015.49. Epub 2015 Apr 7. PMID 25850008
- [Background] Altman KW, Yu GP, Schaefer SD. Consequence of dysphagia in the hospitalized patient: impact on prognosis and hospital resources. Arch Otolaryngol Head Neck Surg. 2010 Aug;136(8):784-9. doi: 10.1001/archoto.2010.129. PMID 20713754
- [Background] Hinchey JA, Shephard T, Furie K, Smith D, Wang D, Tonn S; Stroke Practice Improvement Network Investigators. Formal dysphagia screening protocols prevent pneumonia. Stroke. 2005 Sep;36(9):1972-6. doi: 10.1161/01.STR.0000177529.86868.8d. Epub 2005 Aug 18. PMID 16109909
- [Background] Management of Stroke Rehabilitation Working Group. VA/DOD Clinical practice guideline for the management of stroke rehabilitation. J Rehabil Res Dev. 2010;47(9):1-43. No abstract available. PMID 21213454
- [Background] Donovan NJ, Daniels SK, Edmiaston J, Weinhardt J, Summers D, Mitchell PH; American Heart Association Council on Cardiovascular Nursing and Stroke Council. Dysphagia screening: state of the art: invitational conference proceeding from the State-of-the-Art Nursing Symposium, International Stroke Conference 2012. Stroke. 2013 Apr;44(4):e24-31. doi: 10.1161/STR.0b013e3182877f57. Epub 2013 Feb 14. No abstract available. PMID 23412377
- [Background] O'Horo JC, Rogus-Pulia N, Garcia-Arguello L, Robbins J, Safdar N. Bedside diagnosis of dysphagia: a systematic review. J Hosp Med. 2015 Apr;10(4):256-65. doi: 10.1002/jhm.2313. Epub 2015 Jan 12. PMID 25581840
- [Background] Kertscher B, Speyer R, Palmieri M, Plant C. Bedside screening to detect oropharyngeal dysphagia in patients with neurological disorders: an updated systematic review. Dysphagia. 2014 Apr;29(2):204-12. doi: 10.1007/s00455-013-9490-9. Epub 2013 Sep 13. PMID 24026520
- [Background] Swets JA. The science of choosing the right decision threshold in high-stakes diagnostics. Am Psychol. 1992 Apr;47(4):522-32. doi: 10.1037//0003-066x.47.4.522. PMID 1595983
- [Background] Zammit-Maempel I, Chapple CL, Leslie P. Radiation dose in videofluoroscopic swallow studies. Dysphagia. 2007 Jan;22(1):13-5. doi: 10.1007/s00455-006-9031-x. Epub 2006 Oct 6. PMID 17024550
- [Background] Moro L, Cazzani C. Dynamic swallowing study and radiation dose to patients. Radiol Med. 2006 Feb;111(1):123-9. doi: 10.1007/s11547-006-0013-8. English, Italian. PMID 16623312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was stopped on 23 July 2018 when the announcement of futility stopping was made.
Period: Overall Study
Arm/Group | Single-arm Dysphagia Detection System
Started | 452
Completed | 438
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Single-arm Dysphagia Detection System
Number analyzed (Participants) | 452
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [58 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 286
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 78
  White | 331
  More than one race | 17
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Receiver Operating Characteristic (ROC) Curve to Compare the DDS Predicted Swallow Safety Outcome (Binary) vs. Clinical Reference Standard VFS for THIN-Ba
Description: The primary efficacy of the DDS was measured as the sensitivity & specificity obtained from comparing the DDS predicted swallow safety outcome (binary) with the clinical reference standard VFSS swallow safety outcome (binary) for thin barium (THIN-Ba) stimuli, using 5 boluses per subject protocol. ROC (AUC) was used for comparing the 2 algorithms.
  The ROC curve incorporates both sensitivity (true positive rate) and specificity (true negative rate) providing a single assessment incorporating both measures. The higher the total area under the curve, the greater the predictive power of the outcome.
  Primary analysis for futility was based on 242 subjects (Interim Analysis). The study was terminated based on futility as the AUC for primary endpoint (0.64) was less than the guiding futility bound of 0.75.
Time Frame: The study procedure of simultaneous VFSS and DDS measurement using thin barium (THIN-Ba) was completed in one day for each subject.
Population: The interim analysis data consists of all subjects enrolled and completed before the data cut-off date. The analysis data set consisted of N=253 subjects with N=242 subjects meeting all inclusion-exclusion criteria and having at least one successfully completed Thin bolus swallow measurement (both VFS and DDS).
Measure: Number; unit: Probability
Arm/Group | Single-arm Dysphagia Detection System
Number analyzed (Participants) | 242
Probability | 0.64
Statistical Analysis 1: Comparison: Single-arm Dysphagia Detection System; Test type: Other; AUC under ROC curve = 0.64, 95% CI 1-sided [upper limit 0.72]

2. Secondary Outcome: AUC Under ROC Curve to Compare the DDS Predicted Swallow Safety Outcome (Binary) vs. Clinical Reference Standard VFS for MILD-Ba
Description: The sensitivity & specificity obtained from comparing the DDS predicted swallow safety outcome (binary) with the clinical reference standard VFSS swallow safety outcome (binary) for MILD barium (MILD-Ba) stimuli, using 4 boluses per subject protocol. ROC (AUC) was used for comparing the 2 algorithms. The higher the total AUC, the greater the predictive power of the outcome.
Time Frame: The study procedure of simultaneous VFSS and DDS measurement using mild barium (MILD-Ba) was completed in one day for each subject.
Population: Primary analysis for futility was based on 242 subjects (Interim Analysis).
Measure: Number; unit: Probability
Arm/Group | Single-arm Dysphagia Detection System
Number analyzed (Participants) | 242
Probability | 0.65
Statistical Analysis 1: Comparison: Single-arm Dysphagia Detection System; Test type: Other; AUC under ROC curve = 0.65

3. Secondary Outcome: AUC Under ROC Curve to Compare the DDS Predicted Swallow Safety Outcome (Binary) vs. Clinical Reference Standard VFS for MOD-Ba
Description: The sensitivity & specificity obtained from comparing the DDS predicted swallow safety outcome (binary) with the clinical reference standard VFSS swallow safety outcome (binary) for MODERATE barium (MOD-Ba) stimuli, using 3 boluses per subject protocol. ROC (AUC) was used for comparing the 2 algorithms. The higher the total AUC, the greater the predictive power of the outcome.
Time Frame: The study procedure of simultaneous VFSS and DDS measurement using MOD-Ba was completed in one day for each subject.
Population: Primary analysis for futility was based on 242 subjects (Interim Analysis).
Measure: Number; unit: Probability
Arm/Group | Single-arm Dysphagia Detection System
Number analyzed (Participants) | 242
Probability | 0.576
Statistical Analysis 1: Comparison: Single-arm Dysphagia Detection System; Test type: Other; AUC under ROC curve = 0.576

4. Secondary Outcome: The Sensitivity & Specificity for Swallow Efficiency Using THIN-Ba
Description: The sensitivity & specificity obtained from comparing the DDS predicted swallow efficiency outcome (binary) with the clinical reference standard VFSS swallow efficiency outcome (binary) for Thin barium (THIN-Ba) stimuli.
Time Frame: The study procedure of simultaneous VFSS and DDS measurement using THIN-Ba was completed in one day for each subject.
Population: The analysis for secondary endpoints were to be carried out in a hierarchical fashion in the specified order, only if primary endpoint was met:
  1. swallow safety using MILD-Ba
  2. swallow safety using MOD-Ba
  3. swallow efficiency using THIN-Ba
  4. swallow efficiency using MILD-Ba
  5. swallow efficiency using MOD-Ba
  Outcomes on swallow efficiency were not analyzed.
Arm/Group | Single-arm Dysphagia Detection System
Number analyzed (Participants) | 0

5. Secondary Outcome: The Sensitivity & Specificity for Swallow Efficiency Using MILD-Ba
Description: The sensitivity & specificity obtained from comparing the DDS predicted swallow efficiency outcome (binary) with the clinical reference standard VFSS swallow efficiency outcome (binary) for MILD-Ba.
Time Frame: The study procedure of simultaneous VFSS and DDS measurement using MILD-Ba was completed in one day for each subject.
Population: as for outcome 4
Arm/Group | Single-arm Dysphagia Detection System
Number analyzed (Participants) | 0

6. Secondary Outcome: The Sensitivity & Specificity for Swallow Efficiency Using MOD-Ba
Description: The sensitivity & specificity obtained from comparing the DDS predicted swallow efficiency outcome (binary) with the clinical reference standard VFSS swallow efficiency outcome (binary) for MOD-Ba stimuli.
Time Frame: The study procedure of simultaneous VFSS and DDS measurement using MOD-Ba was completed in one day for each subject.
Population: as for outcome 4
Arm/Group | Single-arm Dysphagia Detection System
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study procedure of simultaneous VFSS and DDS measurement were completed in one day and the subjects were followed for 2 business days after the study procedure to monitor for adverse events.
Groups:
- Dysphagia Detection System (DDS): A trial to test DDS in assessing swallowing safety and efficiency in patients at risk of oropharyngeal dysphagia. Each patient will go through a series of swallows using 5 Thin-BA boluses, 4 Mild-BA boluses and 4 Mod-BA boluses.
Arm/Group | Dysphagia Detection System (DDS)
All-Cause Mortality (participants affected / at risk) | 1/438
Serious Adverse Events (participants affected / at risk) | 5/438
Other Adverse Events (participants affected / at risk) | 0/438
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysphagia Detection System (DDS) (N=438)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Gastrostomy (Surgical and medical procedures) | 2 (2)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT03387267/Prot_002.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03387267/SAP_003.pdf